CLINICAL TRIAL: NCT02043886
Title: The Use of Acarbose to Treat Postprandial Hypotension in Older Adults With Type 2 Diabetes
Brief Title: Acarbose, Postprandial Hypotension and Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Principal Investigator, Kenneth Madden, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H07-00510
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes; Postprandial Hypotension
Keywords: Type 2 Diabetes, Postprandial Hypotension, Acarbose
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acarbose (Active Comparator): Acarbose 50mg by mouth at minute 0 of the Meal Test.
  Interventions: Drug: Acarbose
- Placebo (Placebo Comparator): Placebo 1 tablet at 0 minutes of Meal Test.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acarbose — Acarbose 50 mg by mouth given during Meal Test
  Other Names: Prandase, Precose
  Arms: Acarbose
Drug: Placebo — Non active substance matched to look like Acarbose 50 mg tablets. Taken by mouth during Meal Test.
  Arms: Placebo

SUMMARY:
Postprandial hypotension carries a risk of significant morbidity and morbidity including syncope, falls, dizziness, fatigue, stroke and myocardial infarction. Current therapy consists of dietary manipulation (smaller meals) caffeine and octreotide injections all of which are suboptimal and poorly studied.

The study hypothesis is that administration of Acarbose will decrease the drop in blood pressure and increase in heart rate in response to food in people with Type 2 diabetes.

Acarbose suppresses postprandial glycemia be slowing digestion in the small intestine and delaying gastric emptying.

This is a placebo-controlled cross over study involving 2 - 4 hour Meal Tests. During the meal tests heart rate, blood pressure, cerebral artery velocity will be measured. During one meal test subjects will receive Acarbose 50 mg po and during the other will receive placebo. Order of treatment assignment will be done in randomized fashion. A total of approximately 200 cc of blood will be drawn during each meal test.

ELIGIBILITY:
Inclusion Criteria:

* age 65 year and older
* Type 2 diabetes

Exclusion Criteria:

* less than 65 years of age

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-06; Primary Completion 2013-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Heart rate | continuously during Meal Test; about 4 hours
  Heart rate will be measured continuously by Finometer during the Meal Tests. Each Meal Test will take approximately 4 hours
Blood pressure | Continuously during Meal Tests (approximately 4 hours)
  Blood pressure will be measured continuously by Finometer during each of the Meal Tests (approximately 4 hours)
Middle cerebral artery velocity | continuously during Meal Tests (approximately 4 hours)
  Middle cerebral artery velocity will be measure continuously by transcranial doppler during the Meal Tests (approximately 4 hours)
Serum glucose | Every 15 minutes during Meal Tests
  Serum glucose will be measured using a YSI (Yellow Spring Instruments) Stat 2300 Blood Glucose Analyzer
Serum insulin | Every 15 minutes during Meal Tests (approximately 4 hours)
  Serum insulin levels will be collected every 15 minutes during the Meal Tests (approximately 4 hours) and analyzed by Elisa (enzyme linked immunoabsorbant) assays.
Serum peptides: GIP (gastric inhibitory polypeptide) and GLP-1 (glucagon like peptide) | Every 15 minutes during Meal Tests (approximately 4 hours)
  Serum peptides will be collected every 15 minutes for the duration of the Meal Tests (approximately 4 hours) and analyzed by Elisa (enzyme linked immunoabsorbant) assays.
Catecholamines | Continuously during Meal Test (approximately 4 hours)
  Serum insulin levels will be collected every 15 minutes during the Meal Tests (approximately 4 hours) and analyzed by Elisa (enzyme linked immunoabsorbant) assays.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Madden, MD, Principal Investigator — University of British Columbia
Locations (1):
- VITALiTY Research Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No